CLINICAL TRIAL: NCT01598025
Title: Biparental HLA Haplotype Disparate T-cell Depleted Transplants for Patients Lacking an HLACompatible Donor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to poor accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-053
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Acute Leukemia; Chronic Leukemia; Myelodysplastic Syndrome; Non-Hodgkins Lymphoma
Keywords: ANTITHYMOCYTE GLOBULIN:ATG; FLUDARABINE; THI0TEPA; CliniMACS-CD34 Reagent System; 12-053
MeSH Terms: conditions — Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — Whole-Body Irradiation; Thiotepa; fludarabine phosphate; Melphalan; Antilymphocyte Serum; Peripheral Blood Stem Cell Transplantation

ARMS (2):
- REGIMEN 1 (Experimental): REGIMEN 1: Patients undergo hyperfractionated TBI TID for a total of 11-12 doses on days -10 to -7 and receive thiotepa IV over 4 hours QD on days -6 and -5, fludarabine phosphate IV over 30 minutes QD on days -6 to -2, and anti-thymocyte globulin IV on days -4 to -2.
  TRANSPLANTATION: Patients undergo CD34-selected allogeneic PBSCT on day 0.
  Interventions: Radiation: total-body irradiation (TBI); Drug: thiotepa; Drug: fludarabine phosphate; Biological: anti-thymocyte globulin; Procedure: allogeneic hematopoietic stem cell transplantation; Biological: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis
- Regimen 2 (Experimental): To be given to patients non-malignant, life-threatening diseases and patients with hematologic malignancies, with extensive prior therapy and comorbidities who are unable to receive TBI, consists of Melphalan 70mg/m2 IV x 2 days, thiotepa 5mg/kg IV x 2 days (or 10mg/kg x 1 day), and fludarabine 25 mg/m2 IV x 5 days.
  TRANSPLANTATION: Patients undergo CD34-selected allogeneic PBSCT on day 0.
  Interventions: Drug: thiotepa; Drug: fludarabine phosphate; Drug: melphalan; Biological: anti-thymocyte globulin; Procedure: allogeneic hematopoietic stem cell transplantation; Biological: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: total-body irradiation (TBI)
  Arms: REGIMEN 1
Drug: thiotepa
Drug: fludarabine phosphate
Drug: melphalan
  Arms: Regimen 2
Biological: anti-thymocyte globulin
Procedure: allogeneic hematopoietic stem cell transplantation
Biological: peripheral blood stem cell transplantation
Other: laboratory biomarker analysis

SUMMARY:
Approximately 30% of patients who are candidates for bone marrow transplants do not have an HLA-matched, or close to matched, donor available. For this reason, doctors have been testing ways to make transplants from HLA-partially matched donors as safe and effective as transplants from HLA-matched donors.

This study is being done to test the safety and the treatment results of a specific kind of transplant. In this transplant, blood from two donors will be used. Each donor will share one half of your HLA type. Blood from both donors will be transplanted at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Malignant conditions for which CD34+ selected, T-cell depleted allogeneic hematopoietic stem cell transplantation is indicated such as:

AML in 1st remission - for patients whose AML does not have 'good risk' cytogenetic features (i.e. t 8;21, t15;17, inv 16).

* Secondary AML in 1st remission
* AML in 1st relapse or > 2nd remission
* ALL/LL in 1st remission clinical or molecular features indicating a high risk for relapse; or ALL > 2nd remission
* CML failing to respond to or not tolerating Imatinib, dasatinib, or nilotinib in first chronic phase of disease; or CML in accelerated phase or second chronic phase.
* Non-Hodgkins lymphoma with chemoresponsive disease in any of the following categories: a) intermediate or high grade lymphomas who have failed to achieve a first CR or have relapsed following a 1st remission who are not candidates for autologous transplants.
* any NHL in remission which is considered not curable with chemotherapy alone and not eligible/appropriate for autologous transplant. Myelodysplastic syndrome (MDS): RA/RCMD with high risk cytogenetic features or transfusion dependence, RAEB-1 and RAEB-2 and Acute myelogenous leukemia (AML) evolved from MDS, who are not eligible for transplantation under protocol IRB 08-008.
* Chronic myelomonocytic leukemia: CMML-1 and CMML-2.
* Other rare lethal disorders of Hematopoiesis and Lymphopoiesis for which a T-cell depleted transplant is indicated (e.g. hemophagocytic lymphohistiocytosis; refractory aplastic anemia or conjugated cytopenias; non-SCID lethal genetic immunodeficiencies such as Wiskott Aldrich Syndrome, CD40 ligand deficiency, ALPS).
* Patients may be of either gender and of any racial or ethnic background.
* Patients must have a Karnofsky (adult) or Lansky (pediatric) Performance Status > 70%.
* Patients must have adequate organ function measured by:

Cardiac: asymptomatic or if symptomatic then LVEF at rest must be > 50% and must improve with exercise.

* Hepatic: < 3x ULN ALT and < 2.0x ULN total serum bilirubin, unless there is congenital benign hyperbilirubinemia.
* Renal: serum creatinine <1.2 mg/dl or if serum creatinine is outside the normal range, then CrCl > 40 ml/min (measured or calculated/estimated)
* Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)
* Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Uncontrolled viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV -I/II
* Presence of leukemia in the CNS.

Donor Inclusion Criteria:

* Each donor must meet criteria outlined by institutional policies
* Donor must have adequate peripheral venous catheter access for leukapheresis or must agree to placement of a central catheter.

Donor Exclusion Criteria:

* Evidence of active infection (including urinary tract infection, or upper respiratory tract infection), viral hepatitis exposure (on screening), unless only HBS Ab+ and HBV DNA negative, or serologic evidence of exposure or infection with HIV-I/II or HTLV-I/II
* If donors do not meet institutional guidelines, exclusion will be considered.

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard O'Reilly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- REGIMEN 1: REGIMEN 1: Patients undergo hyperfractionated TBI TID for a total of 11-12 doses on days -10 to -7 and receive thiotepa IV over 4 hours QD on days -6 and -5, fludarabine phosphate IV over 30 minutes QD on days -6 to -2, and anti-thymocyte globulin IV on days -4 to -2.
  TRANSPLANTATION: Patients undergo CD34-selected allogeneic PBSCT on day 0.
  total-body irradiation (TBI)
  thiotepa
  fludarabine phosphate
  anti-thymocyte globulin
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  laboratory biomarker analysis
- Regimen 2: To be given to patients non-malignant, life-threatening diseases and patients with hematologic malignancies, with extensive prior therapy and comorbidities who are unable to receive TBI, consists of Melphalan 70mg/m2 IV x 2 days, thiotepa 5mg/kg IV x 2 days (or 10mg/kg x 1 day), and fludarabine 25 mg/m2 IV x 5 days.
  TRANSPLANTATION: Patients undergo CD34-selected allogeneic PBSCT on day 0.
  thiotepa
  fludarabine phosphate
  melphalan
  anti-thymocyte globulin
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  laboratory biomarker analysis
Period: Overall Study
Arm/Group | REGIMEN 1 | Regimen 2
Started | 0 | 3
Completed | 0 | 0
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: Zero participants were enrolled to Regimen 1
Groups:
- Total: Total of all reporting groups
Arm/Group | REGIMEN 1 | Regimen 2 | Total
Number analyzed (Participants) | 0 | 3 | 3
Age, Continuous [Median (Full Range); unit: years] |  | 12 [11 to 17] | 12 [11 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of HLA-haploidentical Biparental T-cell Depleted CD34+ Peripheral Blood Stem Cell Transplants
Description: Efficacy is measured by:
  1. incidence of transplant-related mortality, overall survival and disease-free survival at 1 year post transplant.
  2. incidence, tempo and complications of engraftment and hematopoietic reconstitutions and conversely, the risk of graft failure
  3. incidence and severity of acute and/or chronic GVHD
  4. incidence and severity of opportunistic infections developing following engraftment
Time Frame: 1 year
Population: Due to the small accrual on study, as well as patient course following treatment on study, the primary objectives of this study were not able to be analyzed.
Arm/Group | REGIMEN 1 | Regimen 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Evaluation of Recipients Post Transplant
Description: The levels of engraftment and persistence of hematopoietic cells and their myeloid and lymphoid progressing from each donor post transplant. The tolerance or reactivity of engrafted T cells from each donor detected in the blood at 3, 6, and thereafter every 3-6 months until normal, post transplant against host cells and cells derived from the other parent as measured by standard mixed lymphocyte culture and cell mediated cytolysis assays.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | REGIMEN 1 | Regimen 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months after transplant
Arm/Group | Regimen 2
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 2 (N=3)
Acidosis (Metabolism and nutrition disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Vascular disorders) | 1
Hypoxia (Reproductive system and breast disorders) | 2
Multi-organ failure (General disorders) | 1
Myelitis (Infections and infestations) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 2 (N=3)
Lymphocyte count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
White blood cell decreased (Investigations) | 3
Anemia (Blood and lymphatic system disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Neutrophil count decreased (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Lipase increased (Investigations) | 1
Serum amylase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT01598025/Prot_SAP_000.pdf